CLINICAL TRIAL: NCT04997655
Title: The Effect of Upper Transabdominal Plain Block on Diaphragm Thickness in Adult Patients After Laparoscopic Cholecystectomy Operation
Brief Title: The Effect of Upper Transabdominal Plain Block on Diaphragm Thickness
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Assoc. Prof. Dr. Yasin Tire, Konya City Hospital
Other Study IDs: KonyaCityH
Record Dates: First submitted 2021-07-25; First posted 2021-08-09 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia, General
Keywords: Laparoscopic Cholecystectomy Operation; Diaphragm Thickness; Upper Transabdominal Plain Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upper Transabdominal Plain Block: All patients in this group are routinely administered general anesthesia. After extubation, the subcostal transverse abdominis area block was directed laterally along the rectus abdominis muscle by finding the linea alba under the xiphoid region under ultrasound guidance with a 22G echogenic block needle, and 20 ml (8 ml 0.5% bupivacaine, 7 ml prilocaine) into the fascia between the rectus abdominis and transverse abdominis muscles. , 5 ml of saline) drug mixture will be performed by the anesthesiologist in charge of that day, who is not aware of the observational measurement to be made, if there is an indication, as a blind practitioner.
  Interventions: Diagnostic Test: Ultrasound measurement
- Opioid analgesia: All patients in this group are routinely administered general anesthesia. Apart from this, in the other group, which does not have peripheral nerve block and only routine opioid analgesia is considered sufficient, only routine peroperative USG diaphragm measurements will be recorded observationally.
  Interventions: Diagnostic Test: Ultrasound measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement — In the patient group who will undergo elective laparoscopic cholecystectomy, the diaphragmatic thickness values measured and recorded routinely at the pre-operative, post-extubation and post-operative 30th minute, at the end of inspiration and expiration, and the inspiratory amplitude in m-mode in the ultrasound measured from the right anterior axillary line subcostal area were observed as observational data. will be saved in our file.

SUMMARY:
In the study, patients of both sexes between the ages of 18 and 60 who will undergo laparoscopic cholecystectomy will be examined. In this patient group, the change in the inspiratory and expiratory diaphragmatic thickness before and after laparoscopic cholecystectomy operation in the upper transabdominal block group will be examined.

DETAILED DESCRIPTION:
The use of ultrasonography (USG) in operating rooms is increasing day by day. Diaphragm thickness can be evaluated by ultrasonography and is used as a bedside method studies have proven that the evaluation of diaphragmatic thickness contributes to the observation of diaphragmatic function and the evaluation of respiratory workload. Measurement of diaphragmatic thickness is a method used in operating rooms and intensive care units to make the decision to wean from mechanical ventilation and extubation. Laparoscopic gallbladder operations are a very common operation in the adult age group in the operating room. In these cases who were intubated and extubated at the end of the operation, regression in respiratory function is observed, especially due to right upper quadrant pain appropriate to the location of the liver. For this reason, the respiratory functions of patients who will have gallbladder surgery will be routinely evaluated before and after gallbladder surgery in our clinic with the help of USG and routinely apply analgesic methods, including peripheral nerve blocks, to patients with pain.

In this study, it will be planned to observe the effect of upper transabdominal area block, which is routinely performed post-operatively in laparoscopic gallbladder operations, on diaphragmatic thickness and therefore on respiratory capacity, and observationally evaluating diaphragmatic thickness measurements by USG, which is routinely performed post-operatively and the measurement records are noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-60
* Both sexes
* Patiets are evaluated as ASA 1 and ASA 2 anesthesia risk, will be examined.

Exclusion Criteria:

* Under 18 years old, over 60 years old
* BMI>35 kg/m2
* Bleeding diathesis
* Local anesthetic allergy
* Infection in the area of TAP (Trans abdominal plane) block application
* Illiteracy, communication problem
* Previous upper abdomen operation
* Transition to open surgery Cases
* Severe chronic respiratory disease
* Neuromuscular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients between the ages of 18-60, of both sexes, who will undergo laparoscopic cholecystectomy, which are evaluated as ASA 1 and ASA 2 anesthesia risk, will be examined.
Study Population: With the calculated sample size values, we will need to include at least 68 patients in our study at 0.5 sensitivity and 0.95 power.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Diaphragm Thickness | 5 minutes before general anesthesia
  The measurement of Diaphragm Thickness by USG
Diaphragm Thickness | 5 minutes after surgery
  The measurement of Diaphragm Thickness by USG
Diaphragm Thickness | 5 minutes after upper abdominal plane block
  The measurement of Diaphragm Thickness by USG

SECONDARY OUTCOMES:
Oxygen saturation | Before the anesthesia, after anesthesia and after 30 minutes in the post operative care unit.
  Oxygen saturation separately for each primary outcome stage
Visual analogue scale | Before the anesthesia, after anesthesia and after 30 minutes in the post operative care unit.
  The patient's pain will be asked in a scale from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Tire, Study Director — Konya City Hospital
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I plan to make individual participant data (IPD) available to only responsible researchers.

REFERENCES:
- [Background] Vivier E, Muller M, Putegnat JB, Steyer J, Barrau S, Boissier F, Bourdin G, Mekontso-Dessap A, Levrat A, Pommier C, Thille AW. Inability of Diaphragm Ultrasound to Predict Extubation Failure: A Multicenter Study. Chest. 2019 Jun;155(6):1131-1139. doi: 10.1016/j.chest.2019.03.004. Epub 2019 Mar 23. PMID 30910636
- [Result] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Result] Dres M, Demoule A. Monitoring diaphragm function in the ICU. Curr Opin Crit Care. 2020 Feb;26(1):18-25. doi: 10.1097/MCC.0000000000000682. PMID 31876624
- See also: Gülleroğlu, Aykan, et al. "Laparoskopik kolesistektomi operasyonlarında karın içi basınç artışının solunum mekaniği, hemodinami ve metabolizma üzerindeki etkileri." Ok Meydanı Eğitim ve Araştırma Hastanesi Anesteziyoloji ve Reanimasyon Kli — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=G%C3%BCllero%C4%9Flu%2C+Aykan%2C+et+al.+%22Laparoskopik+kolesistektomi+operasyonlar%C4%B1nda+kar%C4%B1n+i%C3%A7i+bas%C4%B1n%C3%A7+art%C4%B1%C5%9F%C4%B1n%C4%B1n+solunum+mekani%C4%9Fi%2C+hemodinami+ve+metabolizma+%C3%BCzerindeki+etkileri.%22+Ok+Meydan%C4%B1+E%C4%9Fitim+ve+Ara%C5%9Ft%C4%B1rma+Hastanesi+Anesteziyoloji+ve+Reanimasyon+Klini%C4%9Fi+Uzmanl%C4%B1k+Tezi+%282008%29.&btnG=
- See also: Andıç, K. D., N. Göğüş, and Ayşe Lafcı. "Laparoskopik Kolesistektomi Geçiren Hastalarda Ultrasonografi Eşliğinde Uygulanan Transversus Abdominis Plan Bloğun Perioperatif Analjezi ve Hasta Konforuna Katkısı." (2021). — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=And%C4%B1%C3%A7%2C+K.+D.%2C+N.+G%C3%B6%C4%9F%C3%BC%C5%9F%2C+and+Ay%C5%9Fe+Lafc%C4%B1.+%22Laparoskopik+Kolesistektomi+Ge%C3%A7iren+Hastalarda+Ultrasonografi+E%C5%9Fli%C4%9Finde+Uygulanan+Transversus+Abdominis+Plan+Blo%C4%9Fun+Perioperatif+Analjezi+ve+Hasta+Konforuna+Katk%C4%B1s%C4%B1.%22+%282021%29.&btnG=